CLINICAL TRIAL: NCT05277896
Title: The Randomized Trial of Sedative Choice for Intubation
Brief Title: Randomized Trial of Sedative Choice for Intubation
Acronym: RSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jonathan Casey, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210500; K23HL153584 (NIH); BPS-2022C3-30021 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Failure
Keywords: Critical illness; Emergency airway management; Tracheal intubation; Ketamine; Etomidate
MeSH Terms: conditions — Critical Illness | interventions — Ketamine; Etomidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Active Comparator): Patients in the ketamine group will be assigned to receive intravenous ketamine for induction of anesthesia during tracheal intubation. A dose of 2 mg/kg will be recommended, and the group assignment sheet will contain a nomogram providing the recommended dose for a range of patient weights (in pounds and kg). In this pragmatic trial, treating clinicians will be able elect to give a lesser or greater dose of ketamine than recommended if felt to be required for optimal patient care.
  Interventions: Drug: Ketamine
- Etomidate Group (Active Comparator): Patients in the etomidate group will be assigned to receive intravenous etomidate for induction of anesthesia during tracheal intubation. A dose of 0.3 mg/kg will be recommended, and the group assignment sheet will contain a nomogram providing the recommended dose for a range of patient weights (in pounds and kg). In this pragmatic trial, treating clinicians will be able elect to give a lesser or greater dose of etomidate than recommended if felt to be required for optimal patient care.
  Interventions: Drug: Etomidate

INTERVENTIONS:
Drug: Ketamine — Intravenous ketamine as the sedative for induction of anesthesia during emergency tracheal intubation
  Arms: Ketamine Group
Drug: Etomidate — Intravenous etomidate as the sedative for induction of anesthesia during emergency tracheal intubation
  Arms: Etomidate Group

SUMMARY:
Among critically ill adults undergoing emergency tracheal intubation, one in five experience hypotension, cardiac arrest, or death. The sedatives used to rapidly induce anesthesia for emergency tracheal intubation have been hypothesized to effect cardiovascular complications and patient outcomes, but the optimal sedative medication for intubation of critically ill adults remains unknown. Ketamine and etomidate are the two most commonly used sedatives during intubation of critically ill adults. Data from a randomized clinical trial are urgently needed to determine the effect of ketamine versus etomidate on cardiovascular complications and clinical outcomes of emergency tracheal intubation.

DETAILED DESCRIPTION:
Each year more than 1.5 million critically ill adults receive invasive mechanical ventilation in the United States, at a cost of nearly $30 billion dollars annually. Recent research has dramatically improved patient safety during the maintenance, weaning, and liberation stages of invasive mechanical ventilation. In contrast, the optimal approach to the initiation of mechanical ventilation remains an important knowledge gap in the care of adults with respiratory failure. Among critically ill adults, life-threatening complications during tracheal intubation and initiation of invasive mechanical ventilation remain common. One in five patients experiences hypotension and one-in-forty experiences cardiac arrest during the two-minute tracheal intubation procedure

Cardiovascular collapse is a peri-procedural outcome defined as severe hypotension, new or increased vasopressors, cardiac arrest or death. The occurrence of cardiovascular collapse during tracheal intubation of critically ill adults increases patients' risk of in-hospital mortality. Randomized trials examining intubation technique commonly target cardiovascular collapse as an outcome. Adherence to recommended best-practices for tracheal intubation (e.g., preoxygenation, optimization of patient positioning, and procedural checklists) are insufficient to prevent 20-40% of critically ill adults from experiencing cardiovascular collapse during tracheal intubation.

Rapid sequence induction and tracheal intubation, the most common method of intubation for critically ill patients, is the nearly simultaneous administration of a sedative medication and neuromuscular blocking medication. The ideal sedative agent for rapid sequence intubation would rapidly provide a deep state of unconsciousness and analgesia without causing hemodynamic side effects. No available agent meets all of these criteria. The administration of any of the available sedative agents at a dose large enough to rapidly induce unconsciousness contributes to cardiovascular collapse through vasodilation, decreased cardiac filling pressures from sedation-induced venodilation, and decreased endogenous catecholamines. While all sedatives commonly used during emergency tracheal intubation of critically ill patients have been associated with unsatisfactory hypotension (21 CFR 50.24(a)(1)), ketamine and etomidate are the medications used most commonly in clinical practice due to their rapid onset and favorable hemodynamic profiles relative to the other available sedatives. Other sedatives that have been used in some settings during rapid sequence intubation include benzodiazepines, propofol, and barbiturates. Benzodiazepines do not provide any analgesia and are associated with an unsatisfactory degree of hypotension, with a drop in mean arterial blood pressure of 10 to 25 percent, even among healthy patients. At present, barbiturates are rarely used for tracheal intubation in the US because of unsatisfactorily high rates of post-intubation hypotension and evidence of negative cardiac ionotropy. While propofol is commonly used to induce anesthesia among healthy patients, and is commonly administered as a continuous infusion to maintain sedation for critically ill patients, it is used less commonly as a bolus during tracheal intubation of critically ill patients because it has been suggested to cause unsatisfactorily high rates of hypotension and cardiac depression, compared to ketamine or etomidate.

Ketamine is a phencyclidine derivative that provides anesthesia via its effect at the NMDA receptors. Ketamine has been approved by the United States Food and Drug Administration (FDA) with approved indications including "use as the sole anesthetic agent for diagnostic and surgical procedures that do not require skeletal muscle relaxation" and "induction of anesthesia prior to the administration of other general anesthetic agents." In addition to sedation, ketamine provides significant amnesia and analgesia via action at the opioid receptors, and is commonly used for procedural sedation and as a continuous infusion to control pain.

Ketamine activates the sympathetic nervous system, stimulating the release of catecholamines, which may increase heart rate and blood pressure during intubation and prevent peri-procedural cardiovascular collapse. Conversely ketamine has direct negative ionotropic effects, leading to myocardial depression. While the myocardial depression may be counteracted by increased catecholamine release, ketamine could cause cardiovascular collapse among patients with depleted catecholamine stores, and case reports of unexpected cardiac arrest during intubations with ketamine have been published. Despite stimulating the release of catecholamines, using ketamine as the induction agent during emergency tracheal intubation does not appear to frequently cause or worsen hypertensive urgency or emergency; however, the literature on this topic is limited to case reports.

Historically, concerns have been raised that ketamine might increase intracranial pressure and cause deleterious decreases in cranial perfusion pressure. Recent studies have suggested, however, that ketamine may be associated with a beneficial increase in cranial perfusion pressure as a result of increased mean arterial pressure, and a recent, large before-after study showed no significant differences in clinical outcomes for trauma patients intubated with ketamine versus etomidate.

Etomidate is an imidazole derivative that acts at gamma-aminobutyric acid "A" (GABA) receptors. Etomidate has been approved by the FDA with an indication for "induction of general anesthesia." In a recent review of more than 19,000 intubations by a large, multicenter emergency medicine registry, etomidate was the most commonly used sedative during emergency tracheal intubation.

Etomidate causes less hemodynamic instability than propofol or midazolam, but the data regarding the relative risk of hemodynamical instability with etomidate, compared to ketamine, is unclear. It was initially suggested that ketamine might cause less hypotension than etomidate, given ketamine's ability to stimulate the release of catecholamines, but a recent observational study comparing ketamine and etomidate among nearly 7,000 critically ill adults undergoing tracheal intubation in emergency departments suggested that ketamine was independently associated with an increased risk of peri-intubation hypotension.

Etomidate was initially used both for induction of anesthesia and as a continuous drip for maintenance of anesthesia. Its use as a continuous drip for maintenance of anesthesia was halted after it was discovered that prolonged use of etomidate causes inhibition of adrenal cortisol production by blockade of 11-β-hydroxylase, leading to adrenal insufficiency, and increased mortality. Etomidate use as a single bolus for induction of anesthesia has continued, but numerous studies have demonstrated that even a single dose of etomidate can cause transient adrenal insufficiency. The clinical significance of this relative adrenal insufficiency, however, remains unclear. Contrasting observational studies have suggested that etomidate may have positive, negative or neutral impacts on mortality.

Two randomized trials have directly compared ketamine to etomidate for RSI among critically ill adults. The Ketased trial, published in 2009, was a 469-patient trial conducted across 12 emergency medical services and emergency departments in France. Because many patients were enrolled in the pre-hospital setting without continuous blood pressure monitoring, peri-procedural outcomes such as cardiovascular collapse were not collected, and the results were indeterminate, in regards to the primary outcome, average Sequential Organ Failure Assessment (SOFA) scores in the 72 hours after intubation. The results, however, demonstrated significant heterogeneity. Patients with trauma (for whom increased intracranial pressure from ketamine may be important) experienced a non-significant 4% absolute increase in mortality when intubated with ketamine compared to etomidate. All other patients experienced a non-significantly lower mortality when intubated with ketamine, particularly patients with sepsis who experienced a non-significant 7% absolute mortality benefit (and in whom adrenal insufficiency from etomidate may be particularly important).

The EvK trial, published in January 2022, was a single-center, 801-patient trial conducted among hospitalized patients at a single hospital in Texas.61 Survival at 7 days, the primary outcome of the EvK trial, was higher in the ketamine group, compared to the etomidate group (85.1% vs 77.3%; p=0.005), but this difference was attenuated by day 28, at which point it was no longer significant (66.8% vs 64.1%, p=0.294). The conclusion of this single-center trial was that "there was no significant difference in survival by Day 28", however it was noted that this "could represent a small but durable long-term survival effect, one which our trial was under-powered to detect."

Experts have pointed out that the currently available data on sedative choice during tracheal intubation of critically ill patients are inadequate and have called for additional randomized clinical trials. Because (1) cardiovascular collapse is common during tracheal intubation of critically ill adults (2) sedatives are a driver of cardiovascular collapse, (3) use of ketamine or etomidate varies between centers, specialties, and operators, and (4) prior data suggests the potential for ketamine to significantly decrease mortality for patients without trauma, a large, multicenter trial is needed to determine the effects of ketamine and etomidate on mortality in non-traumatic critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Patient is critically ill and undergoing emergency tracheal intubation with sedation in an enrolling unit
* Planned procedure is orotracheal intubation using a laryngoscope
* Planned operator is a clinician expected to routinely perform tracheal intubation in the participating unit

Exclusion Criteria:

* Patient is known to be less than 18 years old
* Patient is known to be pregnant
* Patient is known to be a prisoner
* Patient is known to have an allergy to ketamine or etomidate
* Patient is presenting to the emergency department with a primary diagnosis of trauma
* Patient or LAR declines participation during pre-enrollment opt-out conversation or by wearing opt-out bracelet for the RSI trial
* Clinician feels ketamine is required or contraindicated for the optimal care of the patient
* Clinician feels etomidate is required or contraindicated for the optimal care of the patient
* Clinician feels an induction medication other than ketamine or etomidate is required for the optimal care of the patient
* Immediate need for intubation precludes safe performance of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2367 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-09-06 (Actual); Study Completion 2025-09-06 (Actual)

PRIMARY OUTCOMES:
All-cause, 28-day, in-hospital mortality | 28 days

SECONDARY OUTCOMES:
Cardiovascular Collapse | from induction to 2 minutes following tracheal intubation
  A composite of any of the following between induction and 2 minutes after intubation:
  * Systolic blood pressure < 65 mmHg
  * New or increased vasopressors
  * Cardiac arrest not resulting in death within 1 hour of induction
  * Cardiac arrest resulting in death within 1 hour of induction

OTHER OUTCOMES:
Cormack-Lehane Grade of glottic view | Duration of procedure (minutes)
  Grade of glottic view on first attempt at intubation:
  Grade 1: Full view of glottis Grade 2: Partial view of glottis Grade 3: Only epiglottis seen (none of glottis) Grade 4: Neither glottis nor epiglottis seen
Time from induction to successful tracheal intubation | Duration of procedure (minutes)
Lowest oxygen saturation between induction and two minutes after intubation | from induction to 2 minutes following tracheal intubation
Lowest oxygen saturation < 80% between induction to two minutes after intubation | from induction to 2 minutes following tracheal intubation
Highest and lowest systolic blood pressure from induction to two minutes after intubation | from induction to 2 minutes following tracheal intubation
Systolic blood pressure > 180 between induction and two minutes after intubation | from induction to 2 minutes following tracheal intubation
Systolic blood pressure < 65 mmHg between induction and 2 minutes after intubation | from induction to 2 minutes following tracheal intubation
New or increased vasopressor between induction and 2 minutes after intubation | from induction to 2 minutes following tracheal intubation
Cardiac arrest within 2 minutes of intubation not resulting in death within 1 hour of induction | from induction to 2 minutes following tracheal intubation
Cardiac arrest within 2 minutes of intubation resulting in death within 1 hour of induction | from induction to 2 minutes following tracheal intubation
Ventilator-free days to study day 28 | 28 days
Vasopressor-free days to study day 28 | 28 days
ICU-free days to study day 28 | 28 days
Systolic blood pressure at 24 hours after induction | 24 hours
Receipt of vasopressors at 24 hours after induction | 24 hours
Cardiac arrest receiving cardiopulmonary resuscitation between induction and hospital discharge | 28 days
Successful intubation on the first attempt | Duration of procedure (minutes)
  Placement of an endotracheal tube in the trachea with a single insertion of a laryngoscope blade into the mouth and EITHER a single insertion of an endotracheal tube into the mouth OR a single insertion of a bougie into the mouth followed by a single insertion of an endotracheal tube over the bougie into the mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Casey, MD, MSc, Principal Investigator — Vanderbilt University Medical Center; Matthew W Semler, MD, MSc, Study Chair — Vanderbilt University Medical Center; Todd W Rice, MD, MSc, Study Director — Vanderbilt University Medical Center; Wesley H Self, MD, MPH, Study Director — Vanderbilt University Medical Center
Locations (6):
- United States (6):
  - UAB Hospital, Birmingham, Alabama
  - University of Colorado Denver, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Following publication, individual patient data will be made available for sharing to researchers with 1) a signed data access agreement, 2) research testing a hypothesis, 3) a protocol that has been approved by an institutional review board, and 4) a proposal that has received approval from the principal investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication. No end date
Access Criteria: 1. a signed data access agreement
  2. research testing a hypothesis
  3. a protocol that has been approved by an institutional review board
  4. a proposal that has received approval from the principal investigator

REFERENCES:
- [Derived] DeMasi SC, Imhoff B, Lewis AA, Seitz KP, Driver BE, Gibbs KW, Ginde AA, Trent SA, Russell DW, Muhs AL, Prekker ME, Gaillard JP, Resnick-Ault D, Stewart LJ, Whitson MR, Van Schaik GWW, Robinson AE, Palakshappa JA, Aggarwal NR, Brainard JC, Douin DJ, Lyle C, Gandotra S, Lacy AJ, Sherlin KC, Carlson GK, Maycee Cain J, Redman B, Higgins C, Withers C, Beach LL, Gould B, McIntosh J, Lloyd BD, Israel TL, Wang L, Rice TW, Self WH, Han JH, Casey JD, Semler MW. Protocol and Statistical Analysis Plan for a Multicenter Randomized Trial of Ketamine vs Etomidate for Emergency Tracheal Intubation. CHEST Crit Care. 2025 Sep;3(3):100177. doi: 10.1016/j.chstcc.2025.100177. Epub 2025 Aug 13. PMID 41472917
- [Derived] Casey JD, Seitz KP, Driver BE, Gibbs KW, Ginde AA, Trent SA, Russell DW, Muhs AL, Prekker ME, Gaillard JP, Resnick-Ault D, Stewart LJ, Whitson MR, DeMasi SC, Robinson AE, Palakshappa JA, Aggarwal NR, Brainard JC, Douin DJ, Marvi TK, Scott BK, Alber SM, Lyle C, Gandotra S, Van Schaik GW, Lacy AJ, Sherlin KC, Erickson HL, Cain JM, Redman B, Beach LL, Gould B, McIntosh J, Lewis AA, Lloyd BD, Israel TL, Imhoff B, Wang L, Spicer AB, Churpek MM, Rice TW, Self WH, Han JH, Semler MW; RSI Investigators and the Pragmatic Critical Care Research Group. Ketamine or Etomidate for Tracheal Intubation of Critically Ill Adults. N Engl J Med. 2025 Dec 9:10.1056/NEJMoa2511420. doi: 10.1056/NEJMoa2511420. Online ahead of print. PMID 41369227
- [Derived] DeMasi SC, Imhoff B, Lewis AA, Seitz KP, Driver BE, Gibbs KW, Ginde AA, Trent SA, Russell DW, Muhs AL, Prekker ME, Gaillard JP, Resnick-Ault D, Stewart LJ, Whitson MR, Van Schaik GWW, Robinson AE, Palakshappa JA, Aggarwal NR, Brainard JC, Douin DJ, Lyle C, Gandotra S, Lacy AJ, Sherlin KC, Carlson GK, Cain JM, Redman B, Higgins C, Withers C, Beach LL, Gould B, McIntosh J, Lloyd BD, Israel TL, Wang L, Rice TW, Self WH, Han JH, Casey JD, Semler MW; RSI investigators and the Pragmatic Critical Care Research Group. Protocol and Statistical Analysis Plan for the Randomized Trial of Sedative Choice for Intubation (RSI). medRxiv [Preprint]. 2025 Jan 18:2025.01.18.25320768. doi: 10.1101/2025.01.18.25320768. PMID 39867415

DOCUMENTS (1):
  • Informed Consent Form (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT05277896/ICF_000.pdf